CLINICAL TRIAL: NCT03704675
Title: Clinical Trial for the Safety, Tolerability, and Pharmacokinetics of TEW-7197 Under Fed or Fasting in Healthy Male Subjects
Brief Title: Effect of Food on the Pharmacokinetics of TEW-7197 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedPacto, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MP-VAC-105
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — vactosertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Fasted->Fed) (Experimental): Group 1 received a single oral dose in a fasting condition in Period 1, followed by a single oral dose after a high-fat diet in Period 2
  Interventions: Drug: TEW-7197
- Group II(Fed->Fasted) (Experimental): Group 2 received a single oral dose after a high-fat diet in Period 1, followed by a single oral in a fasting condition in Period 2
  Interventions: Drug: TEW-7197

INTERVENTIONS:
Drug: TEW-7197 — Administered orally
  Other Names: Vactosertib

SUMMARY:
Participants in this study will receive 200 milligram (mg) TEW-7197 taken at 7days apart. One dose will be given under fasting . The Other dose will be given with a high fat meal. The study will evaluate the effect of a high fat meal on how much of the drug gets into the blood stream. Side effects will be documented. This study will last approximately 2weeks not including screening.

DETAILED DESCRIPTION:
Through screening (D-30 ~ D-1) prior to the first dose of the investigational product, a total of 16 subjects (Group 1: 8 subjects, Group 2: 8 subjects) who were eligible for the inclusion criteria and exclusion criteria were enrolled. This clinical study has a randomized, open, single dose, 2-sequence, 2-period cross-over design and TEW-7197 50 mg x 4 tablets were administered as a single dose in the same individual for 2 periods after fasting or a high fat diet, and each period was repeated with an interval of at least 1 week of wash-out. Pharmacokinetics and safety were evaluated in all subjects according to the planned schedule

ELIGIBILITY:
Inclusion Criteria:

1. Healthy sterile males
2. BMI 18.0kg/m2 - 27.0 kg/m2
3. No congenital or chronic disease and no pathological symptoms or pathological findings
4. Investigator confirm that the subject is eligible through a medical examination (medical history taking ,vital signs, ECG, cardiac ultrasonography, blood science)

Exclusion Criteria:

1. Has pathological symptoms or pathological findings
2. Has a history of disease that may affect the absorption, distribution, metabolism and excretion of a drug
3. SBP>140 or <90 mmhg , DBP>90 or <60mmHg ,Pulse>100
4. No abnormal Clinical Lab findings

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics:Maximum Concentration (Cmax) | Pre-dose through 24 hours post-dose in each period of the. study
  Maximum Concentration (Cmax)
Pharmacokinetics:Area Under the Concentration Curve (AUC) | Pre-dose through 24 hours post-dose in each period of the. study
  Area Under the Concentration Curve (AUC) of TEW-7197

CONTACTS AND LOCATIONS:
Overall Officials: Sunjin Hwang, MD, Study Director — MedPacto, Inc.
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT03704675/Prot_SAP_000.pdf